CLINICAL TRIAL: NCT00477516
Title: Determination of FDF-23 Levels in Non-suppressible PTH Secretion and the Influence of Inflammation on Fetuin A Levels During Hemodialysis Treatment
Brief Title: Association of FGF-23 and Parathyroid Hormone (PTH) in Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James B. Wetmore, MD (Other)
Responsible Party: Sponsor-Investigator, James B. Wetmore, MD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 10571
Record Dates: First submitted 2007-05-21; First posted 2007-05-23 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: exposure to a high-calcium dialysate bath

INTERVENTIONS:
Procedure: exposure to a high-calcium dialysate bath — Subjects are exposed to a high calcium (3.5 mEq/L) dialysate bath for 150 minutes (part 1). At defined timepoints (0, 45, 90, and 150 min) blood is sampled for calcium, PTH, phosphorous, and FGF-23. At another (later) dialysis session (part 2), the process is repeated except that the subjects are exposed to a normal calcium bath (2.5 mEq/L). For each subject, results from part 1 are compared to the results from part 2.

SUMMARY:
The purpose of this study is to determine how levels of this newly-discovered hormone, called FGF-23, changes in the blood in response to a high calcium dialysis bath during a hemodialysis (HD) treatment, and how this relates to changes in the calcium and PTH levels. We are also studying the effects of dialysis and inflammation on the levels of Fetuin A.

We intend to prospectively study a cohort of end stage renal disease (ESRD) patients on hemodialysis in order to determine whether FDF-23 levels independently affect non-suppressible PTH levels. The relationship between Fetuin A and inflammatory markers will also be determined. By dialyzing patients on 3.5 mEq/L calcium dialysate bath, we seek any relationship between ionized calcium, FGF-23 and PTH.

DETAILED DESCRIPTION:
The goal of this study is to ascertain whether there is a regulatory relationship between the novel phosphorus-regulating polypeptide fibroblast growth factor-23 (FGF-23), ionized calcium (iCa), and parathyroid hormone (PTH) levels. In addition, we will determine if there is an inverse relationship between Fetuin A levels and inflammatory markers, interleukin 6 (IL-6) and C-reactive protein (CRP), during a hemodialysis treatment.

All patients participating in this study will be off Zemplar and/or Sensipar for a washout period of approximately 4 weeks as these medications will interfere with the study. Patients will go through one designated research hemodialysis time for a blood draw. Blood draws will be taken during 4 separate intervals at 0, 45, 90 and 150 minutes. At each interval, 4 tubes of blood will be drawn.

There are no further required blood draws once each designated research HD session has been completed. At the conclusion of the designated research HD session, vitamin D analogue (Zemplar®) and/or Cinacalcet (Sensipar®) will be restarted, and the dose will be adjusted to reflect the subject's recent biochemical markers (Ca, Phos, and iPTH).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Chronic Hemodialysis for more than 3 months
* iPTH levels ≥ 300 pg/ml in the absence of therapy: Cinacalcet (Sensipar ®) and/or 1,25 Vitamin analogues (Zemplar®)
* Corrected Ca ≥ 8.4 mg/dl at time of enrollment
* Ability to stay at least 3 hours during hemodialysis treatment

Exclusion Criteria:

* Pediatric Patients (age ≤ 18 years)
* Those unable to give informed consent
* Dialysis treatment for less than 3 months, or pre-emptive kidney transplantation
* Inability to stay more than 3 hours during a single hemodialysis treatment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
change in serum fibroblast growth factor-23 (FGF-23) | 0, 45, 90, and 150 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Peter W. Santos, D.O, Principal Investigator — University of Kansas Medical Center; James B. Wetmore, M.D., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States